CLINICAL TRIAL: NCT00361348
Title: An Open-label, Randomized, 2-part, Parallel Design Study to Characterize the Effect of Heparin on Palifermin Pharmacokinetics and the Effect of Palifermin on Heparin Pharmacodynamics in Healthy Subjects
Brief Title: Palifermin DDI (Drug Drug Interaction)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050137; NCT00964509 (obsolete NCT alias)
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers
Keywords: Palifermin; drug interaction
MeSH Terms: interventions — Fibroblast Growth Factor 7; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Palifermin (Active Comparator): A single 60µg/kg IV bolus dose of palifermin on Day 1 of the treatment period
  Interventions: Drug: Palifermin
- Palifermin + Heparin (Experimental): A single 60µg/kg IV bolus dose of palifermin on Day 1 of the treatment period + unfractionated heparin for a 2 to 3 day heparin titation/maintenance period and continuing through a 3 day treatment period
  Interventions: Drug: Palifermin; Drug: Heparin
- Heparin (Active Comparator): unfractionated heparin for a 2 to 3 day heparin titation/maintenance period and continuing through a 3 day treatment period
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Palifermin
  Other Names: Kepivance
  Arms: Palifermin; Palifermin + Heparin
Drug: Heparin
  Arms: Heparin; Palifermin + Heparin

SUMMARY:
The purpose of this study is to determine if Paliferim interacts with Heparin.

DETAILED DESCRIPTION:
Heparin has been shown to modulate binding of palifermin to the KGF receptor. Therefore, as part of a post-marketing regulatory commitment with the Food and Drug Administration (FDA), the purpose of this study is to characterize the potential pharmacokinetic and pharmacodynamic drug-drug interaction between a continuous IV infusion of heparin and an IV bolus injection of palifermin. If an interaction is observed during co-administration, it is expected that the outcome would be modulation of clearance of palifermin or a change in heparin activity. Although not commonly conducted, the literature describes heparin drug-drug interaction studies conducted in healthy subjects using both subcutaneous (Grimaudo et al,1988; Kroon et al, 1992) and intravenous (Caplain at al, 1999; Noveck & Hubbard, 2004; Spowart et al, 1988) formulations. Based on these experiences, it is appropriate to investigate heparin drug-drug interactions in healthy subjects.

In this study, subjects will receive a single 60 mcg/kg dose of palifermin either as monotherapy or in conjunction with a continuous heparin infusion. The 60 mcg/kg dose of palifermin explored in this study is identical to the current recommended daily dosage for patients with hematologic malignancies who were undergoing autologous PBPC transplantation after receiving total body irradiation and high-dose chemotherapy: 3 consecutive days administered in two cycles with a 5-day non-dosing interval.

ELIGIBILITY:
Inclusion Criteria: - Inclusion: Baseline aPTT values for all subjects must be within normal range. In addition, all subjects must also test negative for occult blood in the stool, have no history of bleeding disorders or no use of aspirin or NSAIDs within 14 days of study Day 1. Exclusion Criteria: - Exclusion: The study will also exclude subjects who have any evidence or history of thrombocytopenia, heparin-induced thrombocytopenia or other contraindications to heparin (e.g., recent surgeries).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45
Dates: Start 2005-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of a continuous intravenous (IV) infusion of unfractionated heparin on the single-dose pharmacokinetics (PK) of palifermin in healthy subjects.

SECONDARY OUTCOMES:
To evaluate the effect (activated partial thromboplastin time, aPTT) of a single dose of palifermin on unfractionated heparin pharmacodynamics [(PD), AUCaPTT, 0-6, AUCaPTT, 0-24].
To evaluate the safety and tolerability of a single 60 µg/kg intravenous dose of palifermin with or without a continuous IV infusion of heparin.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Biovitrum AB (publ)

REFERENCES:
- [Derived] Yang BB, Gillespie B, Smith B, Smith W, Lissmats A, Rudebeck M, Kullenberg T, Olsson B. Pharmacokinetic and pharmacodynamic interactions between palifermin and heparin. J Clin Pharmacol. 2015 Oct;55(10):1109-18. doi: 10.1002/jcph.516. Epub 2015 May 28. PMID 25880826
- See also: FDA-approved Drug Labeling — http://www.kepivance.com/